CLINICAL TRIAL: NCT01234896
Title: Single-dose Nicotine Pharmacokinetics With Four Oral Nicotine Replacement Products. A Study in Healthy Smokers.
Brief Title: Single-dose Nicotine Pharmacokinetics With Four Oral Nicotine Replacement Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NICTDP1080; 2010-021087-15 (EudraCT Number)
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation, Nicotine pharmacokinetics
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine Chewing Gum; Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nicotine Gum 6 (Experimental): 6 mg Nicotine medicated gum
  Interventions: Drug: Nicotine Medicated Gum
- Nicotine Gum 4 (Active Comparator): 4 mg Nicotine Gum
  Interventions: Drug: 4 mg Nicotine Gum
- Nicotine Gum 2 (Active Comparator): 2 mg Nicotine Gum
  Interventions: Drug: 2 mg Nicotine Gum
- Nicotine Lozenge (Active Comparator): 4 mg Nicotine Lozenge
  Interventions: Drug: 4 mg Nicotine Lozenge

INTERVENTIONS:
Drug: Nicotine Medicated Gum — Dosage Form: Gum; Dosage: 6 mg; Frequency: Once; Duration: 30 minutes
  Other Names: Not marketed
  Arms: Nicotine Gum 6
Drug: 4 mg Nicotine Gum — Dosage Form: Gum; Dosage: 4 mg; Frequency: Once; Duration: 30 minutes
  Other Names: Nicorette® Freshfruit gum
  Arms: Nicotine Gum 4
Drug: 2 mg Nicotine Gum — Dosage Form: Gum; Dosage: 2 mg; Frequency: Once; Duration: 30 minutes
  Other Names: Nicorette® Freshfruit gum
  Arms: Nicotine Gum 2
Drug: 4 mg Nicotine Lozenge — Dosage Form: Lozenge; Dosage: 4 mg; Frequency: Once; Duration: until dissolved
  Other Names: NiQuitin™ Mint lozenge
  Arms: Nicotine Lozenge

SUMMARY:
Single-dose nicotine pharmacokinetics with four oral nicotine replacement products. A study in healthy smokers.

DETAILED DESCRIPTION:
Forty-four (44) healthy male or female subjects will be included. Single doses of an experimental Nicotine medicated chewing gum 6 mg and Nicorette® Freshfruit gum 4 mg and 2 mg and NiQuitin™ Mint lozenge 4 mg will be administered in a standardized mode, on four separate treatment visits. Periods without nicotine replacement therapy, each lasting for at least 36 hours, will separate the treatment visits. The subjects will abstain from smoking from 8 pm the evening before each treatment visit and until the end of each visit. Blood for pharmacokinetic analyses will be drawn before, and at 2, 4, 6, 8, 10, 15, 20, 30, 45, and 60 minutes as well as at 1.5, 2, 4, 6, 8, 10, and 12 hours after, product administration. Subjects will be monitored to capture any adverse events that may occur.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, smoking at least 15 cigarettes daily during at least one year preceding inclusion and BMI between 17.5 and 30.0 kilograms per square meter and a total body weight of at least 55.0 kilograms.
* Female participants of child-bearing potential are required to use a medically acceptable means of birth control.
* A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Pregnancy, lactation or intended pregnancy.
* Treatment with an investigational product or donation or loss of blood within 3 month preceding the first dose of study medication.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 12 hours post-dose
  Cmax, which is the maximum observed plasma concentration, measured in nanograms/milliliter (ng/mL)
Area Under the Curve (AUC)(0-t) | 12 hours post-dose
  AUC(0-t), which is the area under the plasma concentration verses time curve from start of drug administration until the time of the last measurable plasma concentration, calculated as hour * nanograms (ng) per milliliter (mL).
AUC (0-∞) | 12 hours post-dose
  AUC (0-∞), which is the area under the plasma concentration-vs.-time curve from start of drug administration until infinity.

SECONDARY OUTCOMES:
AUC(10 min) | 10 minutes post-dose
  AUC(10 min) which is the area under the plasma concentration verses time curve from start of drug administration until 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- McNeil AB Clinical Pharmacology R&D, Lund, Sweden